CLINICAL TRIAL: NCT05205967
Title: REFLECTION: Real World Evidence for Learnings in Early Cancer Detection, a Clinical Practice Learning Program for Galleri®
Brief Title: REFLECTION: A Clinical Practice Learning Program for Galleri®
Status: Active, not recruiting | Type: Observational
Sponsor: GRAIL, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GRAIL-MA-001
Record Dates: First submitted 2021-09-14; First posted 2022-01-25 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Early Detection of Cancer; Cancer
Keywords: Multi-cancer early detection; Cancer screening; Circulating cell-free tumor DNA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received the Galleri® test.
  Interventions: Other: MCED; Other: SOC

INTERVENTIONS:
Other: MCED — Multi-cancer early detection (MCED) test
Other: SOC — Standard of care cancer screening

SUMMARY:
REFLECTION is a multi-center, prospective, non-interventional, cohort study that will enroll approximately 14,000 individuals who have opted to be screened with Galleri®, a blood-based, multi-cancer early detection (MCED) test in routine clinical settings. The purpose of the study is to understand the real-world experience of Galleri® in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Participant has the ability to understand and the willingness to sign a written informed consent form (ICF);
* Participant is at least 22 years old at the time of consent;
* A provider or their designee has ordered the Galleri® test; and
* Participant has the ability to comprehend the participant questionnaires.

Exclusion Criteria:

* There are no exclusions

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll approximately 14,000 participants who meet the defined eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 14633 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
To describe signal detection and cancer detection within and across sites among participants who opt to receive Galleri® in a real world setting. | Up to 12 Months

SECONDARY OUTCOMES:
Galleri®: To assess the feasibility and acceptability of Galleri® from the perspective of participants and patient-reported outcomes (PROs) in a real-world setting. | Up to 12 Months
HCRU: To assess healthcare resource utilization (HCRU) associated with cancer diagnostic workups for participants with signal detected Galleri® test results. | Up to 12 Months

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Vincere Cancer Center, Scottsdale, Arizona
  - Providence, Burbank, California
  - Providence, St. Jude, Fullerton, California
  - Providence, Mission, Mission Viejo, California
  - Providence, Orange County, Orange, California
  - VA Miami Health Care System, Miami, Florida
  - James A. Haley Veterans Hospital (VA Tampa), Tampa, Florida
  - Southeast Louisiana Veterans Health Care System (SLVHCS) (VA New Orleans), New Orleans, Louisiana
  - Boston VA Research Institute (VA Boston), Boston, Massachusetts
  - Providence, Portland, Oregon
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - VA Wilkes Barre Medical Center, Wilkes-Barre, Pennsylvania
  - Carolina Blood and Cancer Care Associate, Lancaster, South Carolina
  - Carolina Blood and Cancer Care Associates, Rock Hill, South Carolina
  - VA Salt Lake City Health Care System (VASLCHCS), Salt Lake City, Utah
  - WVU University Town Centre Family Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kortlever TL, Ferlizza E, Lauriola M, Borrelli F, Porro A, Spaander MCW, Bossuyt PM, Ricciardiello L, Dekker E. Diagnostic Accuracy of an Add-On, Blood-Based Screening Test for Colorectal Cancer in Two Established Screening Programmes. Aliment Pharmacol Ther. 2025 Jun;61(12):1935-1943. doi: 10.1111/apt.70141. Epub 2025 Apr 10. PMID 40207404